CLINICAL TRIAL: NCT05384860
Title: Incorporating Acupuncture Into ERAS for Ambulatory Total Hip Replacement (THR) Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital for Special Surgery, New York (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2021-1496
Record Dates: First submitted 2022-05-05; First posted 2022-05-20 (Actual); Last update posted 2025-12-11 (Actual); Status verified 2025-02

CONDITIONS: Acupuncture; Hip Surgery; Opioid Use
Keywords: hip surgery; acupuncture
MeSH Terms: interventions — Acupuncture Therapy

STUDY DESIGN:
Intervention Model Description: Subjects were randomly assigned to receive Acupuncture, or No Acupuncture based on a 1:1 schedule with blocks of four created prior to study initiation using SAS version 9.4 (SAS Institute; Cary, NC) by a member of the biostatistics core not otherwise involved in the trial.
  Treatment assignments were transcribed onto notecards and sealed in opaque, consecutively numbered envelopes by a research assistant not otherwise involved in the trial.
  After patient consent and prior to anesthesia start, the research assistant involved in the trial handed the randomization envelope to the medical acupuncturist. All patients and research assistants involved with data collection will be blinded to the group allocation.
  Randomization lists will be accessed by an intra-op monitor RA who is not otherwise involved in the study in any other aspect.
Who Masked: Participant, Outcomes Assessor
Masking Description: Both patients and research assistants (RAs)collecting data from the patients will be blinded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Active Acupuncture Group (Active Comparator): For the patients randomized to the acupuncture group, once sedation has been deemed adequate by the anesthesiologist, a certified medical acupuncturist will perform ipsilateral Auricular Trauma Protocol (ATP) acupuncture at eight ear points (Hypothalamus, Amygdala, Hippocampus, Prefrontal Cortex, Point Zero, Shen Men, Insula, Vagus) with 30Hz electrostimulation at two of those points (Shen Men and Hypothalamus). Acupuncture needles will be left in place and stimulated for 60 min and then removed.
  Interventions: Device: Auricular Trauma Protocol (ATP) Acupuncture
- Placebo No Acupuncture Group (Placebo Comparator): These patients will not receive acupuncture treatment during surgery, their surgery will continue as normal.
  Interventions: Other: No Acupuncture Group

INTERVENTIONS:
Device: Auricular Trauma Protocol (ATP) Acupuncture — Small filiform (needle) like needles use low frequency electrostimulation at eight ear points for 60 minutes while patient is sedated during surgery. All other aspects of the surgical procedure will go as planned according to the hospital's standard of care.
  Arms: Active Acupuncture Group
Other: No Acupuncture Group — This involves not receiving the acupuncture treatment and surgery going entirely as normal according to the hospital's standard of care.
  Arms: Placebo No Acupuncture Group

SUMMARY:
At this time, no formal ERAS (enhanced recovery after surgery) protocol exists for THR that incorporates perioperative acupuncture. Developing, and more importantly, validating a preliminary fast-track protocol for THR can have a significant impact on reducing recovery time and improving the rate at which this subgroup of surgeries is done on an outpatient basis. Furthermore, previous studies of acupuncture as an adjunctive therapy for postoperative analgesia have primarily investigated patient satisfaction rather than the impact on postoperative opioid consumption.

The majority of studies also place acupuncture needles preoperatively, rather than following induction of anesthesia (intra-operatively). This study hopes to show that placing auricular therapy needles intraoperatively is a feasible part of a protocol for motivated patients to minimize opioids after total knee arthroplasty. The prospect of incorporating intraoperative acupuncture as an adjunct into said protocol is very attractive given its low cost, its safety profile, its ease of administration, and the growing evidence supporting its efficacy. This study would provide further clarity on whether perioperative acupuncture can effectively reduce hospital length of stay and post-operative opioid consumption, in addition to evaluating the role of perioperative acupuncture in improving recovery after THR as part of a multimodal fast-track protocol.

ELIGIBILITY:
Inclusion Criteria:

* ASA status of 1 or 2
* Ages 18-80
* Undergoing a total hip replacement
* Ability to follow study protocol
* English-speaking

Exclusion Criteria:

* Non-English speaking
* Chronic opioids use (6 weeks or more)
* Contraindication to neuraxial anesthesia or peripheral nerve block
* Intending to receive general anesthesia
* Contraindication to intra-op protocol
* Implanted cardiac device (i.e. pacemaker)
* Active ear infection
* Non-native ear, previous scarring or surgery
* Ear gauges or other deforming ear piercing
* Allergy to Nickel

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 484 (Actual)
Dates: Start 2022-07-06 (Actual); Primary Completion 2025-04-04 (Actual); Study Completion 2025-04-04 (Actual)

PRIMARY OUTCOMES:
Opioid Usage | Day 30
  The primary outcome is the incidence of patients who maintain a low-dose opioid regimen (71.5 OME or less) out to 30 days post-op. Patient intake of opioid medication will be measured up to the 30 days post-operation.

SECONDARY OUTCOMES:
NRS Pain Scores | Post-operatively in: PACU (post-anesthesia care unit) immediately post-operation, Day 1, Day 2, Day 14 & Day 30
  NRS pain scores at rest and with movement
Satisfaction with Protocol | Day 30
  Satisfaction with the whole protocol/study experience and pain management throughout surgery and recovery. Patients will be asked to rate their satisfaction with the study, care provided and pain management on a scale of 1-10 with 1 being least satisfied and 10 being most satisfied.
Post-operative Nausea & Vomiting (PONV) | Post-operatively in: PACU (post-anesthesia care unit), Day 1
  Incidence of nausea, vomiting, pruritus, constipation
Range of Motion | Post-operatively on: Day 1 and Day 14
  Postoperative range of motion (extension and flexion)
Pain Catastrophizing Scale (PCS) | Pre-operative
  13-item self-report measure designed to assess catastrophic thinking related to pain among adults with or without chronic pain. It is a self-reported measure with items scored from 0-4 with 4 being the most catastrophic. The higher a patient's total scores the more catastrophic their thoughts are in relation to pain.
Center for Epidemiologic Studies Short Depression Scale & Anxiety Scale (CES-D) | Pre-operative
  20 questions that asks about various symptoms of depression as they have occurred in the past week. Response options range from 0 to 3 for each item (0 = Rarely or None of the Time, 1 = Some or Little of the Time, 2 = Moderately or Much of the time, 3 = Most or Almost All the Time). Total scores range from 0 to 60, with higher scores indicated greater depressive symptoms.
Hours to Discharge | Will be assessed up to 4 days post-operatively or until patient leaves hospital.
  The total number of hours patients spend in the hospital until discharge from the hospital. This will be measured from the start of surgery in the OR until discharge from hospital.

CONTACTS AND LOCATIONS:
Overall Officials: Stephanie Cheng, MD, Principal Investigator — Hospital for Special Surgery, New York
Locations (1):
- Hospital for Special Surgery, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in this article after de-identification (text, tables, figures, and appendices).
Supporting Information: Study Protocol
Time Frame: Beginning 9 months and ending 36 months following article publication.
Access Criteria: Investigators whose proposed use of the data has been approved by an Independent review committee ("learned intermediary") identified for this purpose and who have signed a DUA.